CLINICAL TRIAL: NCT03460002
Title: A Cluster Randomized Controlled Trial on the Campaign Effect of Measles Vaccine and Oral Polio Vaccine on General Hospital Admissions and Mortality Among Children
Brief Title: Vaccine Campaign Effects on General Hospital Admissions and Mortality Among Children
Acronym: RE-CAMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Statens Serum Institut (Other); Research Center for Vitamins and Vaccines (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RE-CAMP
Record Dates: First submitted 2016-11-21; First posted 2018-03-09 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Measles Vaccination; Oral Polio Vaccine; Non-specific/Heterologous Effects of Vaccines; Mortality; Morbidity; Children
Keywords: Measles vaccine; Oral polio vaccine; Campaign; Child mortality; Child morbidity; Non-specific effects
MeSH Terms: interventions — Measles Vaccine; Poliovirus Vaccine, Oral

STUDY DESIGN:
Intervention Model Description: The RECAMP trials test two separate hypotheses relating to the potential beneficial non-specific effects of providing live vaccines in general vaccination campaigns.
  The RECAMP-MV trial tests the effect of a Measles Vaccination campaign among children aged 9-59 months The RECAMP-OPV trial tests the effect of an Oral Polio Vaccination campaign in children aged 0-8 months
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Measles vaccine (Experimental): In intervention villages children will be weighed and receive standard measles vaccine in one dose if they are between 9-59 months old.
  Interventions: Biological: Measles vaccine
- Oral polio vaccine (Experimental): In intervention villages children will be weighed and receive standard oral polio vaccine in one or two doses if they are between 0-8 months old.
  Interventions: Biological: Oral polio vaccine
- Weighing-MV (No Intervention): In control villages children aged 9-59 months acting as controls to the MV-intervention arm will be weighed only.
- Weighing-OPV (No Intervention): In control villages children aged 0-8 months acting as controls to the OPV-intervention arm will be weighed only.

INTERVENTIONS:
Biological: Measles vaccine — A measles vaccine prequalified from the World Health Organization will be administered in one dose by deep subcutaneous injection into the left subscapular region by a local nurse.
  Arms: Measles vaccine
Biological: Oral polio vaccine — A bivalent oral polio vaccine prequalified by the World Health Organization will be administered in one or two doses directly into the mouth of the vaccinee with two drops per dose by a local nurse.
  Arms: Oral polio vaccine

SUMMARY:
The world is set on eradicating measles and polio infections in the coming decade. Once both infections are under control, campaigns with measles and oral polio vaccines will be phased out. This might do more harm than good for child survival in low-income countries. Studies from the Bandim Health Project in Guinea-Bissau, and elsewhere, have revealed, that the live measles and oral polio vaccines have beneficial non-specific effects, i.e. effects on child morbidity and mortality unrelated to prevention of the targeted diseases.

The campaigns are presumed to be most beneficial for children not reached by routine vaccination programs, as they are not already protected. However, studies show that prior routine or campaign vaccination may boost resistance against unrelated infections. If we phase out measles and oral polio campaigns after eradicating their target infections without considering the impact on child survival, the drastic decline in child mortality since 1990 could change direction. We will conduct the first cluster randomized controlled trial to evaluate the effect of measles and oral polio campaigns on general child morbidity and mortality via the Bandim Health Project. Bandim Health Project runs a Health and Demographic Surveillance System in Guinea-Bissau since 1978 and assesses child health interventions' real-life effects, via continuous registration of all interventions given to all children, and follow-up of individuals. We will conduct the trials in rural Guinea-Bissau monitoring all nine health regions.

The hypotheses are:

RECAMP-MV: Measles vaccination campaign in Guinea-Bissau reduce morbidity and mortality among children between 9 and 59 months of age by 80% during the subsequent 18 months in a context of limited measles infection.

RECAMP-OPV: Oral polio vaccination campaigns in Guinea-Bissau reduce morbidity and mortality among children between 0 and 8 months of age by 25% during the subsequent 12 months in a context with no polio infection.

Originally, the trials were meant to be implemented in 182 clusters, enrolling 21000 children. Following revised sample size calculations and discussions with the Data Safety and Monitoring Board, the number of clusters were increased to 222 and the planned number of enrolments increased from 21,000 to 28,000 (RECAMP-MV: 18000, RECAMP-OPV: 10000).

To explore the hypothesis that at least part of the beneficial non-specific effects of OPV is driven by changes in the gut and/or respiratory microbiome, we will collect microbiome samples in a sub-group:

A nasal swab and a rectal swab will be collected from 50 infants allocated to the intervention group, and 50 infants allocated to the control group. Two sample will be collected for each infant one when recruited for RECAMP-OPV and a second two months later.

ELIGIBILITY:
Inclusion Criteria: Children aged 0-59 months living with families registered in the rural Bandim Health Project Health and Demographic Surveillance Site are included, provided a parent/guardian consent.

Exclusion Criteria:

* the child has temperature > 39.0◦C or a severe acute illness as defined by the examining nurse

OR

* the child has as a mid upper arm circumference < 110 mm and is older than 6 months (most feasible local indicator of AIDS and chronic immunosuppressive disease)

OR

* the child has experienced a severe allergic reaction after previous vaccination, drug or food.

OR

* the child is enrolled in an ongoing study of Bacillus Calmette Guerin vaccine and is < 2 months old

OR

* For the RECAMP-MV trial: the child is enrolled in RECAMP-OPV

Ages: 0 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28612 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Composite outcome: mortality and hospital admission (measured as a rate) | Enrolment to end of study (longest follow-up 2 years)
  Death (registered through follow-up visits, verified by verbal autopsies) or first admission (overnight stay at hospital registered by interview at follow up visits)
  Correction: Non-accidental death (registered through follow-up visits, verified by verbal autopsies) or first admission not caused by accident (overnight stay at hospital registered by interview at follow up visits) The outcomes were correctly specified in the protocol paper and analysis plan (doi: 10.1186/s12889-019-7813-y)

SECONDARY OUTCOMES:
Nutritional status | Enrolment to end of study (longest follow-up 2 years)
  Mid-upper-arm-circumference registered with measurement tape as per UNICEF recommendations
Mortality | Enrolment to end of study (longest follow-up 2 years)
  Death (registered through follow-up visits, verified by verbal autopsies)
  Corrections: Non-accidental death (registered through follow-up visits, verified by verbal autopsies) The outcome was correctly specified in the protocol paper and analysis plan (doi: 10.1186/s12889-019-7813-y)
Hospital admission | Enrolment to end of study (longest follow-up 2 years)
  admission (overnight stay at hospital registered by interview at follow up visits)
  Correction: admission not caused by accident (overnight stay at hospital registered by interview at follow up visits) The outcome was correctly specified in the protocol paper and analysis plan (doi: 10.1186/s12889-019-7813-y)

OTHER OUTCOMES:
Acute adverse reactions | One-two months after a child is included in the study
  Health center consultations and illness registered through follow-up visits
Changes to the Respiratory and Gut Microbiome | Two months after a child is included in the study
  Among 100 children enrolled in the OPV or corresponding control arm (Weighing-OPV), a nasal swab and a rectal swab will be collected at enrolment and 2 months later to assess effects of campaign OPV on the microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Ane Fisker, MD, PhD, Principal Investigator — Bandim Health Project, Guinea-Bissau and Statens Serum Institute, Research Center for Vitamins and Vaccines, Bandim Health Project; Peter Aaby, DMSc,Professor, Principal Investigator — Bandim Health Project, Guinea-Bissau and Statens Serum Institute, Research Center for Vitamins and Vaccines, Bandim Health Project; Aksel Jensen, PhD, Principal Investigator — Statens Serum Institute, Research Center for Vitamins and Vaccines, Bandim Health Project; Anshu Varma, MSc, Principal Investigator — Statens Serum Institute, Research Center for Vitamins and Vaccines, Bandim Health Project; Amabelia Rodrigues, Ph, Principal Investigator — Bandim Health Project, Guinea-Bissau
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] World Health Organization. Global measles and rubella strategic plan: 2012-2020. 2012.
- [Background] World Health Organization. Polio eradication and endgame strategic plan: 2013-2018. 2013.
- [Background] Meeting of the Strategic Advisory Group of Experts on immunization, October 2015 - conclusions and recommendations. Wkly Epidemiol Rec. 2015 Dec 11;90(50):681-99. No abstract available. English, French. PMID 26685390
- [Background] Kristensen I, Aaby P, Jensen H. Routine vaccinations and child survival: follow up study in Guinea-Bissau, West Africa. BMJ. 2000 Dec 9;321(7274):1435-8. doi: 10.1136/bmj.321.7274.1435. PMID 11110734
- [Background] Aaby P, Samb B, Simondon F, Seck AM, Knudsen K, Whittle H. Non-specific beneficial effect of measles immunisation: analysis of mortality studies from developing countries. BMJ. 1995 Aug 19;311(7003):481-5. doi: 10.1136/bmj.311.7003.481. PMID 7647643
- [Background] Aaby P, Garly ML, Bale C, Martins C, Jensen H, Lisse I, Whittle H. Survival of previously measles-vaccinated and measles-unvaccinated children in an emergency situation: an unplanned study. Pediatr Infect Dis J. 2003 Sep;22(9):798-805. doi: 10.1097/01.inf.0000083821.33187.b5. PMID 14506371
- [Background] Aaby P, Martins CL, Garly ML, Bale C, Andersen A, Rodrigues A, Ravn H, Lisse IM, Benn CS, Whittle HC. Non-specific effects of standard measles vaccine at 4.5 and 9 months of age on childhood mortality: randomised controlled trial. BMJ. 2010 Nov 30;341:c6495. doi: 10.1136/bmj.c6495. PMID 21118875
- [Background] Lund N, Andersen A, Hansen AS, Jepsen FS, Barbosa A, Biering-Sorensen S, Rodrigues A, Ravn H, Aaby P, Benn CS. The Effect of Oral Polio Vaccine at Birth on Infant Mortality: A Randomized Trial. Clin Infect Dis. 2015 Nov 15;61(10):1504-11. doi: 10.1093/cid/civ617. Epub 2015 Jul 28. PMID 26219694
- [Background] Lund N, Biering-Sorensen S, Andersen A, Monteiro I, Camala L, Jorgensen MJ, Aaby P, Benn CS. Neonatal vitamin A supplementation associated with a cluster of deaths and poor early growth in a randomised trial among low-birth-weight boys of vitamin A versus oral polio vaccine at birth. BMC Pediatr. 2014 Aug 28;14:214. doi: 10.1186/1471-2431-14-214. PMID 25163399
- [Background] Martins CL, Benn CS, Andersen A, Bale C, Schaltz-Buchholzer F, Do VA, Rodrigues A, Aaby P, Ravn H, Whittle H, Garly ML. A randomized trial of a standard dose of Edmonston-Zagreb measles vaccine given at 4.5 months of age: effect on total hospital admissions. J Infect Dis. 2014 Jun 1;209(11):1731-8. doi: 10.1093/infdis/jit804. Epub 2014 Jan 16. PMID 24436454
- [Background] Sorup S, Benn CS, Poulsen A, Krause TG, Aaby P, Ravn H. Live vaccine against measles, mumps, and rubella and the risk of hospital admissions for nontargeted infections. JAMA. 2014 Feb 26;311(8):826-35. doi: 10.1001/jama.2014.470. PMID 24570246
- [Background] Sorup S, Stensballe LG, Krause TG, Aaby P, Benn CS, Ravn H. Oral Polio Vaccination and Hospital Admissions With Non-Polio Infections in Denmark: Nationwide Retrospective Cohort Study. Open Forum Infect Dis. 2015 Dec 17;3(1):ofv204. doi: 10.1093/ofid/ofv204. eCollection 2016 Jan. PMID 26885538
- [Background] Aaby P, Hedegaard K, Sodemann M, Nhante E, Veirum JE, Jakobsen M, Lisse I, Jensen H, Sandstrom A. Childhood mortality after oral polio immunisation campaign in Guinea-Bissau. Vaccine. 2005 Feb 25;23(14):1746-51. doi: 10.1016/j.vaccine.2004.02.054. PMID 15705481
- [Background] Andersen A, Fisker AB, Rodrigues A, et al. National immunization campaigns with oral polio vaccine (OPV) reduce the general all-cause mortality rate: An analysis of the effect of campaign-OPV on child mortality within seven randomised trials (submitted). 2016.
- [Background] Fisker AB, Rodrigues A, Martins C, Ravn H, Byberg S, Thysen S, Storgaard L, Pedersen M, Fernandes M, Benn CS, Aaby P. Reduced All-cause Child Mortality After General Measles Vaccination Campaign in Rural Guinea-Bissau. Pediatr Infect Dis J. 2015 Dec;34(12):1369-76. doi: 10.1097/INF.0000000000000896. PMID 26379164
- [Background] Benn CS, Netea MG, Selin LK, Aaby P. A small jab - a big effect: nonspecific immunomodulation by vaccines. Trends Immunol. 2013 Sep;34(9):431-9. doi: 10.1016/j.it.2013.04.004. Epub 2013 May 14. PMID 23680130
- [Background] Byberg S, Thysen SM, Rodrigues A, Martins C, Cabral C, Careme M, Aaby P, Benn CS, Fisker AB. A general measles vaccination campaign in urban Guinea-Bissau: Comparing child mortality among participants and non-participants. Vaccine. 2017 Jan 3;35(1):33-39. doi: 10.1016/j.vaccine.2016.11.049. Epub 2016 Nov 24. PMID 27890397
- [Background] Aaby P, Andersen M, Sodemann M, Jakobsen M, Gomes J, Fernandes M. Reduced childhood mortality after standard measles vaccination at 4-8 months compared with 9-11 months of age. BMJ. 1993 Nov 20;307(6915):1308-11. doi: 10.1136/bmj.307.6915.1308. PMID 8257884
- [Background] World Bank. World Bank Countries and Lending Groups. https://datahelpdesk.worldbank.org/knowledgebase/articles/906519 (accessed 01-07-2016).
- [Background] United Nations Inter-agency Group for Child Mortality Estimation. http://www.childmortality.org/index.php?r=site/graph#ID=GNB_Guinea-Bissau (accessed 01-07-2016)
- [Background] INDEPTH network. Indepth Verbal Autopsy. http://www.indepth-network.org/resources/tools (accessed 25-07-2016).
- [Background] Desgrees du Lou A, Pison G, Aaby P. Role of immunizations in the recent decline in childhood mortality and the changes in the female/male mortality ratio in rural Senegal. Am J Epidemiol. 1995 Sep 15;142(6):643-52. doi: 10.1093/oxfordjournals.aje.a117688. PMID 7653475
- [Background] Aaby P, Jensen H, Samb B, Cisse B, Sodemann M, Jakobsen M, Poulsen A, Rodrigues A, Lisse IM, Simondon F, Whittle H. Differences in female-male mortality after high-titre measles vaccine and association with subsequent vaccination with diphtheria-tetanus-pertussis and inactivated poliovirus: reanalysis of West African studies. Lancet. 2003 Jun 28;361(9376):2183-8. doi: 10.1016/S0140-6736(03)13771-3. PMID 12842371
- [Background] Benn CS, Rodrigues A, Yazdanbakhsh M, Fisker AB, Ravn H, Whittle H, Aaby P. The effect of high-dose vitamin A supplementation administered with BCG vaccine at birth may be modified by subsequent DTP vaccination. Vaccine. 2009 May 11;27(21):2891-8. doi: 10.1016/j.vaccine.2009.02.080. Epub 2009 Mar 9. PMID 19428899
- [Background] Benn CS, Fisker AB, Whittle HC, Aaby P. Revaccination with Live Attenuated Vaccines Confer Additional Beneficial Nonspecific Effects on Overall Survival: A Review. EBioMedicine. 2016 Aug;10:312-7. doi: 10.1016/j.ebiom.2016.07.016. Epub 2016 Jul 15. PMID 27498365
- [Background] World Health Organization. Information Sheet Observed Rate of Vaccine Reactions Measles, Mumps and Rubella Vaccines. 2014. http://www.who.int/vaccine_safety/initiative/tools/MMR_vaccine_rates_ information_sheet.pdf (accessed 01-07-2016).
- [Background] World Health Organization. Information Sheet Observed Rate of Vaccine Reactions Polio Vaccines. 2014. http://www.who.int/vaccine_safety/initiative/tools/Polio_vaccine_rates_information_sheet.pdf (accessed 01-07-2016).
- [Background] Chuang SK, Lau YL, Lim WL, Chow CB, Tsang T, Tse LY. Mass measles immunization campaign: experience in the Hong Kong Special Administrative Region of China. Bull World Health Organ. 2002;80(7):585-91. Epub 2002 Jul 30. PMID 12163924
- [Background] Abedi GR, Mutuc JD, Lawler J, Leroy ZC, Hudson JM, Blog DS, Schulte CR, Rausch-Phung E, Ogbuanu IU, Gallagher K, Kutty PK. Adverse events following a third dose of measles, mumps, and rubella vaccine in a mumps outbreak. Vaccine. 2012 Nov 19;30(49):7052-8. doi: 10.1016/j.vaccine.2012.09.053. Epub 2012 Oct 3. PMID 23041123
- [Background] Arruda WO, Kondageski C. Aseptic meningitis in a large MMR vaccine campaign (590,609 people) in Curitiba, Parana, Brazil, 1998. Rev Inst Med Trop Sao Paulo. 2001 Sep-Oct;43(5):301-2. doi: 10.1590/s0036-46652001000500012. PMID 11696855
- [Background] Roberts RJ, Sandifer QD, Evans MR, Nolan-Farrell MZ, Davis PM. Reasons for non-uptake of measles, mumps, and rubella catch up immunisation in a measles epidemic and side effects of the vaccine. BMJ. 1995 Jun 24;310(6995):1629-32. doi: 10.1136/bmj.310.6995.1629. PMID 7795447
- [Background] Strebel PM, Papania MJ, Dayan GH, Halsey NA. Measles Vaccine. In: Plotkin SA, Orenstein WA, Offit PA, eds. Vaccines: Saunders; 2008: 353-98.
- [Background] Fisker AB, Bale C, Jorgensen MJ, Balde I, Hornshoj L, Bibby BM, Aaby P, Benn CS. High-dose vitamin A supplementation administered with vaccinations after 6 months of age: sex-differential adverse reactions and morbidity. Vaccine. 2013 Jun 28;31(31):3191-8. doi: 10.1016/j.vaccine.2013.04.072. Epub 2013 May 14. PMID 23680441
- [Background] Sugawara T, Ohsuka Y, Taya K, Yasui Y, Wada N, Sakano M, Koshida R, Fujii F, Shibata S, Hashimoto G, Utsumi H, Sumitomo M, Ishihara M, Kondo H, Sato H, Ueno K, Araki K, Okabe N. Diarrhea as a minor adverse effect due to oral polio vaccine. Jpn J Infect Dis. 2009 Jan;62(1):51-3. PMID 19168959
- [Background] Meeting of the Strategic Advisory Group of Experts on immunization, April 2013 - conclusions and recommendations. Wkly Epidemiol Rec. 2013 May 17;88(20):201-6. No abstract available. English, French. PMID 23696983
- [Background] Higgins JPT, Soares-Weiser K, Reingold A. Systematic review of the non-specific effects of BCG, DTP and measles containing vaccines . Available at: http://www.who.int/immunization/sage/meetings /2014/april/3_NSE_Epidemiology_review_Report_to_SAGE_14_Mar_FINAL.pdf?ua=1, 2014.
- [Background] Meeting of the Strategic Advisory Group of Experts on immunization, April 2014 -- conclusions and recommendations. Wkly Epidemiol Rec. 2014 May 23;89(21):221-36. No abstract available. English, French. PMID 24864348
- [Background] Aaby P, Gustafson P, Roth A, Rodrigues A, Fernandes M, Sodemann M, Holmgren B, Benn CS, Garly ML, Lisse IM, Jensen H. Vaccinia scars associated with better survival for adults. An observational study from Guinea-Bissau. Vaccine. 2006 Jul 17;24(29-30):5718-25. doi: 10.1016/j.vaccine.2006.04.045. Epub 2006 May 6. PMID 16720061
- [Background] Jensen ML, Dave S, Schim van der Loeff M, da Costa C, Vincent T, Leligdowicz A, Benn CS, Roth A, Ravn H, Lisse IM, Whittle H, Aaby P. Vaccinia scars associated with improved survival among adults in rural Guinea-Bissau. PLoS One. 2006 Dec 20;1(1):e101. doi: 10.1371/journal.pone.0000101. PMID 17183634
- [Background] Rieckmann A, Villumsen M, Sorup S, Haugaard LK, Ravn H, Roth A, Baker JL, Benn CS, Aaby P. Vaccinations against smallpox and tuberculosis are associated with better long-term survival: a Danish case-cohort study 1971-2010. Int J Epidemiol. 2017 Apr 1;46(2):695-705. doi: 10.1093/ije/dyw120. PMID 27380797
- [Derived] Varma A, Aaby P, Thysen SM, Jensen AKG, Fisker AB. Reduction in Short-term Outpatient Consultations After a Campaign With Measles Vaccine in Children Aged 9-59 Months: Substudy Within a Cluster-Randomized Trial. J Pediatric Infect Dis Soc. 2020 Nov 10;9(5):535-543. doi: 10.1093/jpids/piaa091. PMID 32897359
- [Derived] Varma A, Jensen AKG, Thysen SM, Pedersen LM, Aaby P, Fisker AB. Research protocol of two concurrent cluster-randomized trials: Real-life Effect of a CAMPaign with Measles Vaccination (RECAMP-MV) and Real-life Effect of a CAMPaign with Oral Polio Vaccination (RECAMP-OPV) on mortality and morbidity among children in rural Guinea-Bissau. BMC Public Health. 2019 Nov 11;19(1):1506. doi: 10.1186/s12889-019-7813-y. PMID 31711464